CLINICAL TRIAL: NCT07004907
Title: Efficacy and Tolerability of the APD Treatment of Toddlers and Newborns With the Silencia PD Cycler
Brief Title: Efficacy and Tolerability of the APD Treatment in PAED Patients
Acronym: SilenciaPAED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-Silencia-02-LA
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Renal Failure Acute Chronic
Keywords: Automated peritoneal dialysis; paedriatic patients; Kt/V; ultrafiltration; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SilenciaPAED (Experimental): Patients will receive treatment as prescribed by the physician using the Silencia PD cycler.
  Interventions: Device: Treatment with the pedriatic mode of the APD cycler

INTERVENTIONS:
Device: Treatment with the pedriatic mode of the APD cycler — Patients weighing less than 20 kg will be treated for 4 weeks with APD using the PAED mode of the Silencia PD cycler

SUMMARY:
The Silencia PD (peritoneal dialysis) cycler offers a pediatric (PAED) mode with advanced features such as Time and Volume Optimization (TAVO), supporting precise and individualized treatment. This study evaluates the efficacy and tolerability of Automated Peritoneal Dialysis (APD) using the Silencia PD cycler in patients weighing ≤ 20 kg and able to tolerate a minimum inflow volume of 100 mL. The primary objective is to determine whether patients achieve a total weekly Kt/Vurea ≥ 1.8.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by legal representative and investigator/authorized physician
* The minors have received the information referred to in Article 63(2) MDR in a way adapted to their age and mental maturity and from investigators or members of the investigating team who are trained or experienced in working with children
* The explicit wish of a minor who is capable of forming an opinion and assessing the information referred to in Article 63(2) MDR to refuse participation in, or to withdraw from, the clinical investigation at any time, is respected by the investigator
* patients with renal failure treated or planned to be treated with APD
* Body weight ≤ 20 kg
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Any conditions which could interfere with the patient's ability to comply with the study
* Patient or legal representative is not able to give informed consent according to European Medical Device Regulation and corresponding national regulations
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study
* Life expectancy < 3 months
* Patients who suffer from peritonitis/exit site infection during the last 4 weeks

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Total weekly Kt/V urea | The primary endpoint is total Kt/Vurea at week 2 and 4
  The primary objective is to determine whether patients achieve a total weekly Kt/V urea ≥ 1.8.

SECONDARY OUTCOMES:
Mean daily ultrafiltration (UF) | Mean UF will be measured at weeks 2 and 4
Residual renal function (RRF) | RRF will be measured at weeks 2 and 4
  Renal urea clearance
Residual renal function (RRF) | RRF will be measured at weeks 2 and 4
  Renal creatinine clearance
Residual renal function (RRF) | RRF will be measured at weeks 2 and 4
  24h urine output
Residual renal function (RRF) | RRF will be measured at weeks 2 and 4
  GFR (calculated during the analysis)

IPD SHARING:
Plan to Share IPD: No